CLINICAL TRIAL: NCT05827107
Title: A Single-centre, Exploratory Study to Characterise the Skin Barrier and Microbiome of Patients With Cutaneous T-cell Lymphoma (CTCL)
Brief Title: Skin Barrier and Microbiome of CTCL Patients
Status: Completed | Type: Observational
Sponsor: Centre for Human Drug Research, Netherlands (Other)
Collaborators: Leiden University Medical Center (Other); Micreos (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHDR2230
Record Dates: First submitted 2023-03-29; First posted 2023-04-24 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma, T-Cell, Cutaneous
Keywords: CTCL; Microbiome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this study is to investigate the microbiome composition of the nares, non-lesional skin and patches, plaques and tumours in lesional skin of CTCL patients, including all stages of the disease, and to correlate microbiome (including S. aureus presence) and disease severity from CTCL patients.

DETAILED DESCRIPTION:
Cutaneous T-cell lymphomas (CTCL) are primary T-cell derived cutaneous lymphomas; they represent a group of lymphoproliferative disorders characterized by localization of neoplastic T lymphocytes to the skin. This may result in skin patches and plaques, erythroderma, itch, dry skin and hair loss. In advanced stages tumours in the skin occur often associated with cutaneous and systemic infections. Mycosis fungoides (MF), which is generally indolent in behaviour, and Sézary syndrome (SS), an aggressive and leukemic variant, comprise approximately 53% of all primary cutaneous lymphomas and two-third of CTCL (Willemze et al., 2019). Staphylococcus aureus (S. aureus) and its toxins have been shown to positively correlate with progression and colonize 31% to 76% of patients across all stages and subtypes (Fujii, 2021). Staging and diagnosing the progression of CTCL are key to defining an effective treatment strategy. Current treatment strategies for CTCL are diverse, focusing on anti-tumour activity and infection and/or rash treatment.

CTCL is a group of malignancies that is a subset of non-Hodgkin lymphomas derived from skin-homing T cells with no evidence of extracutaneous disease at the time of diagnosis. MF and SS are the most common CTCL variants (Bastidas Torres et al., 2018; Willemze et al., 2019). MF is the most prevalent (up to 60%) clinical form of CTCL and is characterized by proliferation of malignant skin-homing T cells in a chronic inflammatory environment in the skin. SS is a rare - approx. 2% - leukemic type of CTCL, traditionally defined by the triad of pruritic erythroderma, generalized lymphadenopathy, and clonally related neoplastic T cells with cerebriform nuclei (Sézary cells) in the skin, lymph nodes, and peripheral blood (Girardi et al., 2004; Willemze et al., 2019). CTCL shows, besides MF and SS, several other subtypes and presents in several stages of severity.

The skin barrier of CTCL was observed to be perturbed and hypothetically this influences the microbiome - host interaction.

Only limited information is available about the relationship between CTCL variants, its staging, clinical symptoms and S. aureus colonization. In addition, studies assessed mostly S. aureus presence solely, and not the whole microbiome. This study is set up to investigate the microbiological properties of CTCL patients. Furthermore, the microbiome-host interaction will be studied by investigating skin barrier properties and patient-reported aspects in these patients.

This will provide the rationale and potential impact for a subsequent trial assessing the safety and efficacy of a novel topical compound. It will help determine the population eligible for such study, as well as enriching the population with those most likely to benefit from this therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide a written informed consent prior to any study procedures.
2. Male or female subjects, 18 years or older.
3. A confirmed diagnosis of CTCL (MF type or SS type) and stage classification via histology or clinico-histopathological correlation.
4. For the stage IA-IIA CTCL patients: at least one patch and/or one plaque lesion are present, with at least one dimension with a diameter of ≥3 cm. For the stage IIB and higher classified CTCL patients: at least one tumour is present, with at least one dimension with a diameter of ≥1.5 cm.

Exclusion Criteria:

1. Use of topical antibiotic (on selected target lesions) and/or oral antibiotic therapy in the previous 14 days before the visit.
2. Clinically significant skin disease on the selected lesions, other than CTCL or CTCL associated secondary impetiginisation, as judged by the investigator.
3. Ongoing active skin infection, other than secondary impetiginized CTCL lesions.
4. Treatment of selected target CTCL lesions with radiotherapy within 8 weeks prior to Day 1.
5. Any other clinical condition that may preclude participation in the study as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Mycosis fungoides and Sézary syndrome of all stages will be recruited via the patient out clinic for cutaneous lymphoma in the Leiden University Medical Centre.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Microbiome composition of skin lesions (target lesions, nares and non-lesional skin) | baseline visit
Bacterial colonisation via semi-quantitative bacterial culture samples for S. aureus | baseline visit
Correlation of microbiome and culture results with clinical CTCL symptoms and their intra- and inter-patient variability. | baseline visit

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rissmann, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided